CLINICAL TRIAL: NCT00490711
Title: Phase II Study of Sequential Therapy With Paclitaxel Plus Carboplatin Followed by Gemzar Plus Carboplatin in the Treatment of Patients With Epithelial Ovarian Cancer FIGO Stages III-IV
Brief Title: Treatment of Paclitaxel Plus Carboplatin Followed by Gemcitabine Plus Carboplatin for Patients With Epithelial Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4720; B9E-MC-S205
Record Dates: First submitted 2007-06-21; First posted 2007-06-25 (Estimated); Last update posted 2007-06-25 (Estimated); Status verified 2007-06

CONDITIONS: Epithelial Ovarian Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — Gemcitabine; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: gemcitabine
Drug: carboplatin
Drug: paclitaxel

SUMMARY:
The purpose of this study is to evaluate the efficacy of paclitaxel and carboplatin followed by gemcitabine and carboplatin therapy for patients with epithelial ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified epithelial ovarian cancer
* FIGO stage III-IV
* Patients with measurable disease. RECIST criteria with GCIG modifications will be used for response and for progression assessment.
* Lesions serving as measurable disease must have the longest diameter of greater than or equal to 20 mm as measured with conventional techniques or greater than or equal to 10 mm with spiral CT scan. Lesions measured by physical examination must have a longest diameter of greater than or equal to 20 mm.

Exclusion Criteria:

* Ovarian tumors with low malignant potential (borderline tumors)
* Non-epithelial ovarian or mixed epithelial. non epithelial tumors (e.g. mixed Mullerian tumors)
* Time between definitive surgery and enrollment into the study is greater than 6 weeks
* Patients who have received previous chemotherapy or radiotherapy

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2003-07; Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Overall response rate

SECONDARY OUTCOMES:
Progression-free survival
2-year survival
Toxicity
Dose intensity

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bratislava, Slovakia

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com